CLINICAL TRIAL: NCT01255995
Title: The Natural History of Artificial Intraocular Lenses (IOL) in Eyes With Exfoliation Syndrome
Brief Title: Natural History of IOL in Pseudo Exfoliation Syndrome
Acronym: PXF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Other Study IDs: 2PR2240936
Record Dates: First submitted 2010-12-02; First posted 2010-12-08 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Pseudo Exfoliation Syndrome
Keywords: PXF
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Patients: Controls without PXF who require cataract surgery
- Pseudo Exfoliation patients: PXF subjects with or without glaucoma who require cataract surgery
  Interventions: Device: Capsular Tension Ring

INTERVENTIONS:
Device: Capsular Tension Ring — Capsular Tension Ring
  Other Names: CTR
  Groups: Pseudo Exfoliation patients

SUMMARY:
* The purpose of this study is to determine the natural course of IOL in PXF,
* To demonstrate use of a clinical grading system for PXF,
* To strategize a way to prevent IOL dislocation, subluxation post operatively,
* To demonstrate intraoperative and long-term post-operative complications associated with phaco and PXF
* To suggest evidence-based ways to minimize these complications, by using capsular tension rings (CTR), specific IOL material or size

DETAILED DESCRIPTION:
Pseudo exfoliation syndrome (PXF) is a generalized degenerative microfibrillopathy that primarily is manifested with deposits of exfoliative material present on the anterior capsule of the crystalline lens, zonules, papillary margin of the iris, corneal endothelium, ciliary body and the trabecular meshwork. The build of this exfoliative material causes microscopic changes of the zonules and their attachments, causing a weakening of the zonules. These clinical findings have implications not only for cataract surgery, as association of lens opacities with exfoliation syndrome is well documented but also for glaucoma, with exfoliative glaucoma being the most common cause for secondary open angle glaucoma in the world.In patients with exfoliation syndrome, small pupil and phacodonesis, comparison between extra capsular cataract extraction and small incision cataract surgery revealed better best corrected visual acuity and fewer intra and post operative complications with the smaller incision for phacoemulsification. The capsular tension rings (CTR) implanted prior to phacoemulsification reduced intraoperative zonular dialysis, increased the rate of capsular IOL fixation, and improved uncorrected visual acuity. Either the degree of lens change the stage of PXF, or the type of IOL might influence long term outcome in PXF associated with cataract surgery:The postoperative course of those with either more advanced cataract or with more advanced PXF may be different than those who have surgery with less cataract our and/or degree of PXF. The stage of PXF alone at the time of cataract surgery may influence outcome. Once PXF identified, surgery performed at an earlier stage of cataract with a softer lens in XFS results in fewer long term problems following phacoemulsification. A standardized way of clinically measuring/monitoring XFS is helpful during large clinical studies Specific intraocular lens design should be considered when scheduling phacoemulsification in patients with PXF.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75
* PXF with or without secondary open-angle glaucoma who present with cataract and willing to undergo phacoemulsification with IOL
* Nuclear sclerosis with LOCS III grade and above
* Pupil size more than 4mm on dilatation
* Endothelial cell count >1,500
* No visible phacodonesis

Exclusion Criteria:

* Uncontrolled IOP/glaucoma
* History of narrow angles, chronic narrow angle glaucoma
* Any pre-existing clinical zonular dialysis or phacodonesis
* Pseudo uveitis
* One eyed patients
* Cardiac pathology
* Uncontrolled diabetes, hypertension & severe asthma
* Obviously debilitated patients
* Traumatic cataract
* Complicated cataract
* Congenital cataract
* Drug induced cataract
* Shallow anterior Chamber
* Amblyopia
* Dense posterior polar cataract
* Corneal pathology
* Retinal pathology
* RAPD
* Severe visual field defect (MD->12.0dB)
* Diabetic retinopathy
* Combined Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PXF subjects with or without glaucoma who require cataract surgery. Controls without PXF who require cataract surgery
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-12; Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
IOL Centration / IOL Stability | 10th Year

SECONDARY OUTCOMES:
Visual Acuity | 10th Year
Anterior capsular fibrosis/phimosis | 10th Year
New onset of phacodonesis | 10th Year
Development or worsening of glaucoma | 10th Year

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Aravind, MS, Principal Investigator — Aravind Eye Hospital
Locations (4):
- India (4):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu
  - Aravind Eye Hospital, Tirunelveli, Tamil Nadu